CLINICAL TRIAL: NCT03145181
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation Study of Teclistamab, a Humanized BCMA x CD3 Bispecific Antibody in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Dose Escalation Study of Teclistamab, a Humanized BCMA*CD3 Bispecific Antibody, in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: MajesTEC-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108206; 64007957MMY1001 (Other: Janssen Research & Development, LLC); 2016-002122-36 (EudraCT Number); 2023-503438-40-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05463939 (Approved for marketing)
Record Dates: First submitted 2017-04-28; First posted 2017-05-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation (IV) (Experimental): Participants will receive Teclistamab intravenously (IV).
  Interventions: Drug: Teclistamab (IV)
- Part 2: Dose Expansion (IV) (Experimental): Participants will receive Teclistamab IV.
  Interventions: Drug: Teclistamab (IV)
- Part 1: Dose Escalation (SC) (Experimental): Participants will receive Teclistamab subcutaneously (SC).
  Interventions: Drug: Teclistamab(SC)
- Part 2: Dose Expansion (SC) (Experimental): Participants will receive Teclistamab SC.
  Interventions: Drug: Teclistamab(SC)

INTERVENTIONS:
Drug: Teclistamab (IV) — Participants will receive IV infusion of Teclistamab.
  Other Names: JNJ-64007957
  Arms: Part 1: Dose Escalation (IV); Part 2: Dose Expansion (IV)
Drug: Teclistamab(SC) — Participants will receive SC injection of Teclistamab.
  Other Names: JNJ-64007957
  Arms: Part 1: Dose Escalation (SC); Part 2: Dose Expansion (SC)

SUMMARY:
The purpose of this study is to identify the recommended Phase 2 dose(s) (RP2Ds) and schedule assessed to be safe for Teclistamab and to characterize the safety and tolerability of Teclistamab at the RP2Ds.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts, separately for IV and SC administration: dose escalation (Part 1) and dose expansion (Part 2). It will evaluate safety, tolerability, pharmacokinetics and preliminary antitumor activity of Teclistamab administered to adult participants with relapsed or refractory multiple myeloma. The overall safety of the study drug will be assessed by physical examinations, Eastern Cooperative Oncology Group performance status, laboratory tests, vital signs, electrocardiograms, adverse event monitoring, and concomitant medication usage. Disease evaluations will include peripheral blood and bone marrow assessments at screening (performed within 28 days) and to confirm stringent complete response (sCR), complete response (CR), or relapse from CR. The end of study (study completion) is defined as 2 years after the last participant in Part 3 has received his or her initial dose of teclistamab. Study record NCT04557098 is Phase 2 part of this study and study record NCT03145181 is Phase 1 part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Measurable multiple myeloma that is relapsed or refractory to established therapies with known clinical benefit in relapsed/refractory multiple myeloma or be intolerant of those established multiple myeloma therapies, and a candidate for Teclistamab treatment in the opinion of the treating physician. Prior lines of therapy must include a proteasome inhibitor, an immunomodulatory drug and anti-CD38 monoclonal antibody in any order during the course of treatment. Participants who could not tolerate a proteasome inhibitor or immunomodulatory drugs and an anti-CD38 monoclonal antibody are allowed
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Female participants of childbearing potential must use acceptable method of contraception
* Participants must sign an ICF indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study. Consent is to be obtained prior to the initiation of any study-related tests or procedures that are not part of standard-of-care for the participant's disease

Exclusion Criteria:

* Prior treatment with any B cell maturation antigen (BCMA) targeted therapy
* Prior antitumor therapy as follows, before the first dose of study drug: Targeted therapy, epigenetic therapy, or treatment with an investigational drug or used an invasive investigational medical device within 21 days or at least 5 half-lives, whichever is less; Monoclonal antibody treatment for multiple myeloma within 21 days; Cytotoxic therapy within 21 days; Proteasome inhibitor therapy within 14 days; Immunomodulatory agent therapy within 7 days; Gene modified adoptive cell therapy (example, chimeric antigen receptor modified T cells, natural killer [NK] cells) within 3 months; Radiotherapy within 14 days or focal radiation within 7 days
* Toxicities from previous anticancer therapies that have not resolved to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy
* Received a cumulative dose of corticosteroids equivalent to >= 140 milligram (mg) of prednisone within the 14-day period before the first dose of study drug (does not include pretreatment medication)
* Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2027-05-28 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to Day 28
  The Dose Limiting Toxicities (DLTs) are based on drug related adverse events and defined as any of the following events: hematological / non hematological toxicity of Grade 3 or higher.
Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 7 years and 3 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

SECONDARY OUTCOMES:
Teclistamab Serum Concentrations | Up to 8 weeks
  Concentration assessment will be done to evaluate the effect of Teclistamab.
Number of Participants with Teclistamab Antibodies | Up to 8 weeks
  Antibodies to Teclistamab will be assessed to evaluate potential immunogenicity.
Preliminary Antitumor Activity of Teclistamab at the RP2D(s) in Part 2 | Up to End of Treatment (Approximately 91 days)
  Preliminary antitumor activity of Teclistamab will be done using the International Myeloma Working Group (IMWG) response criteria.
Biomarker Assessment | Up to 8 weeks
  Biomarker assessment may be done to evaluate the effect of Teclistamab.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- United States (5):
  - City of Hope, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Icahn School of Medicine at Mount Sinai Program for the Protection of Human Subjects, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
- France (2):
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHRU Tours Hopital Bretonneau, Tours
- VU Medisch Centrum, Amsterdam, Netherlands
- Spain (4):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
- Haematology Centre, R 51, Stockholm, Sweden

REFERENCES:
- [Derived] Martin TG, Mateos MV, Yi JH, van de Donk NWCJ, Cai Z, Fu W, Garfall AL, Iida S, Jung SH, Kuroda Y, Niu T, Nooka AK, Min CK, Sidana S, Chastain K, Doyle M, Nishikawa K, Wang X, Song Y, Yamazaki H, Izumi Y, Zhuo J, Zhu A, Yoon DH, Du J, Ishida T. Efficacy and safety of teclistamab in triple-class exposed relapsed/refractory multiple myeloma: Pooled findings from three clinical cohorts and a retrospective cohort. Cancer. 2026 Jan 1;132(1):e70237. doi: 10.1002/cncr.70237. PMID 41485109
- [Derived] Guo Y, Niu J, Carde NAQ, Wu L, Miao X, Hanson S, Su Y, Ruixo CP, Vishwamitra D, Chastain K, Samtani MN, Wang W, Haddish-Berhane N. Teclistamab Dosing in Responders: Modeling and Simulation Results from the MajesTEC-1 Study in Relapsed/Refractory Multiple Myeloma. Target Oncol. 2025 Jul;20(4):651-661. doi: 10.1007/s11523-025-01149-1. Epub 2025 May 7. PMID 40332715
- [Derived] Touzeau C, Krishnan AY, Moreau P, Perrot A, Usmani SZ, Manier S, Cavo M, Martinez Chamorro C, Nooka AK, Martin TG, Karlin L, Leleu X, Bahlis NJ, Besemer B, Pei L, Stein S, Wang Lin SX, Trancucci D, Verona RI, Girgis S, Miao X, Uhlar CM, Chastain K, Garfall AL. Efficacy and safety of teclistamab in patients with relapsed/refractory multiple myeloma after BCMA-targeting therapies. Blood. 2024 Dec 5;144(23):2375-2388. doi: 10.1182/blood.2023023616. PMID 39172760
- [Derived] Moreau P, Mateos MV, Gonzalez Garcia ME, Einsele H, De Stefano V, Karlin L, Lindsey-Hill J, Besemer B, Vincent L, Kirkpatrick S, Delforge M, Perrot A, van de Donk NWCJ, Pawlyn C, Manier S, Leleu X, Martinez-Lopez J, Ghilotti F, Diels J, Morano R, Albrecht C, Strulev V, Haddad I, Pei L, Kobos R, Smit J, Slavcev M, Marshall A, Weisel K. Comparative Effectiveness of Teclistamab Versus Real-World Physician's Choice of Therapy in LocoMMotion and MoMMent in Triple-Class Exposed Relapsed/Refractory Multiple Myeloma. Adv Ther. 2024 Feb;41(2):696-715. doi: 10.1007/s12325-023-02738-0. Epub 2023 Dec 19. PMID 38110653
- [Derived] Martin TG, Moreau P, Usmani SZ, Garfall A, Mateos MV, San-Miguel JF, Oriol A, Nooka AK, Rosinol L, Chari A, Karlin L, Krishnan A, Bahlis N, Popat R, Besemer B, Martinez-Lopez J, Delforge M, Trancucci D, Pei L, Kobos R, Fastenau J, Gries KS, van de Donk NWCJ. Teclistamab Improves Patient-Reported Symptoms and Health-Related Quality of Life in Relapsed or Refractory Multiple Myeloma: Results From the Phase II MajesTEC-1 Study. Clin Lymphoma Myeloma Leuk. 2024 Mar;24(3):194-202. doi: 10.1016/j.clml.2023.11.001. Epub 2023 Nov 14. PMID 38052709
- [Derived] Nooka AK, Rodriguez C, Mateos MV, Manier S, Chastain K, Banerjee A, Kobos R, Qi K, Verona R, Doyle M, Martin TG, van de Donk NWCJ. Incidence, timing, and management of infections in patients receiving teclistamab for the treatment of relapsed/refractory multiple myeloma in the MajesTEC-1 study. Cancer. 2024 Mar 15;130(6):886-900. doi: 10.1002/cncr.35107. Epub 2023 Nov 14. PMID 37960969
- [Derived] Miao X, Wu LS, Lin SXW, Xu Y, Chen Y, Iwaki Y, Kobos R, Stephenson T, Kemmerer K, Uhlar CM, Banerjee A, Goldberg JD, Trancucci D, Apte A, Verona R, Pei L, Desai R, Hickey K, Su Y, Ouellet D, Samtani MN, Guo Y, Garfall AL, Krishnan A, Usmani SZ, Zhou H, Girgis S. Population Pharmacokinetics and Exposure-Response with Teclistamab in Patients With Relapsed/Refractory Multiple Myeloma: Results From MajesTEC-1. Target Oncol. 2023 Sep;18(5):667-684. doi: 10.1007/s11523-023-00989-z. Epub 2023 Sep 15. PMID 37713090
- [Derived] Moreau P, van de Donk NW, Nahi H, Oriol A, Nooka AK, Martin T, Rosinol L, Karlin L, Benboubker L, Mateos MV, Popat R, Martinez-Lopez J, Sidana S, Delforge M, Pei L, Trancucci D, Olyslager Y, Uhlar C, Stephenson T, Rampelbergh RV, Banerjee A, Kobos R, Usmani SZ. Plain language summary of the MajesTEC-1 study of teclistamab for the treatment of people with relapsed or refractory multiple myeloma. Future Oncol. 2023 Apr;19(12):811-818. doi: 10.2217/fon-2023-0171. Epub 2023 May 3. PMID 37132225
- [Derived] Martin TG, Mateos MV, Nooka A, Banerjee A, Kobos R, Pei L, Qi M, Verona R, Doyle M, Smit J, Sun W, Trancucci D, Uhlar C, van de Donk NWCJ, Rodriguez C. Detailed overview of incidence and management of cytokine release syndrome observed with teclistamab in the MajesTEC-1 study of patients with relapsed/refractory multiple myeloma. Cancer. 2023 Jul 1;129(13):2035-2046. doi: 10.1002/cncr.34756. Epub 2023 Mar 29. PMID 36991547
- [Derived] Girgis S, Lin SXW, Pillarisetti K, Banerjee A, Stephenson T, Ma X, Shetty S, Yang TY, Hilder BW, Jiao Q, Hanna B, Adams HC 3rd, Sun YN, Sharma A, Smit J, Infante JR, Goldberg JD, Elsayed Y. Translational Modeling Predicts Efficacious Therapeutic Dosing Range of Teclistamab for Multiple Myeloma. Target Oncol. 2022 Jul;17(4):433-439. doi: 10.1007/s11523-022-00893-y. Epub 2022 Jun 24. PMID 35749004
- [Derived] Moreau P, Garfall AL, van de Donk NWCJ, Nahi H, San-Miguel JF, Oriol A, Nooka AK, Martin T, Rosinol L, Chari A, Karlin L, Benboubker L, Mateos MV, Bahlis N, Popat R, Besemer B, Martinez-Lopez J, Sidana S, Delforge M, Pei L, Trancucci D, Verona R, Girgis S, Lin SXW, Olyslager Y, Jaffe M, Uhlar C, Stephenson T, Van Rampelbergh R, Banerjee A, Goldberg JD, Kobos R, Krishnan A, Usmani SZ. Teclistamab in Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2022 Aug 11;387(6):495-505. doi: 10.1056/NEJMoa2203478. Epub 2022 Jun 5. PMID 35661166
- [Derived] Usmani SZ, Garfall AL, van de Donk NWCJ, Nahi H, San-Miguel JF, Oriol A, Rosinol L, Chari A, Bhutani M, Karlin L, Benboubker L, Pei L, Verona R, Girgis S, Stephenson T, Elsayed Y, Infante J, Goldberg JD, Banerjee A, Mateos MV, Krishnan A. Teclistamab, a B-cell maturation antigen x CD3 bispecific antibody, in patients with relapsed or refractory multiple myeloma (MajesTEC-1): a multicentre, open-label, single-arm, phase 1 study. Lancet. 2021 Aug 21;398(10301):665-674. doi: 10.1016/S0140-6736(21)01338-6. Epub 2021 Aug 10. PMID 34388396
- [Derived] Pillarisetti K, Powers G, Luistro L, Babich A, Baldwin E, Li Y, Zhang X, Mendonca M, Majewski N, Nanjunda R, Chin D, Packman K, Elsayed Y, Attar R, Gaudet F. Teclistamab is an active T cell-redirecting bispecific antibody against B-cell maturation antigen for multiple myeloma. Blood Adv. 2020 Sep 22;4(18):4538-4549. doi: 10.1182/bloodadvances.2020002393. PMID 32956453
- See also: A Study of Teclistamab, in Participants With Relapsed or Refractory Multiple Myeloma — https://clinicaltrials.gov/ct2/show/NCT04557098